CLINICAL TRIAL: NCT04990128
Title: Randomized Trial on the Evaluation of the Effectiveness of One Single Bone Marrow Aspirate Hip Injection Versus Triamcinolone for Hip Osteoarthritis
Brief Title: Bone Marrow Aspirate Concentrate Versus Triamcinolone Injection For Hip Osteoarthritis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Lisa Dean Moseley Foundation (Unknown)
Responsible Party: Principal Investigator, LEONARDO OLIVEIRA, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLA 21-020; IDE 27066 (Other: FDA)
Record Dates: First submitted 2021-06-22; First posted 2021-08-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hip Osteoarthritis
Keywords: bone marrow aspirate concentrate; triamcinolone
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: bone marrow aspirate concentrate versus triamcinolone
Who Masked: Participant
Masking Description: Participant will undergo a sham bone needling if assigned to Triamcinolone group to keep patient blinded to their intervention. This will simulate the bone marrow aspiration process.
  Outcomes assessor will receive de-identified data including the treatment type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bone marrow aspirate concentrate (Experimental): Bone marrow that is aspirated then concentrated using a device.
  Interventions: Combination Product: Aspire Needle + Emcyte PureBMC
- Triamcinolone (Active Comparator): Triamcinolone is a corticosteroid.
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Combination Product: Aspire Needle + Emcyte PureBMC — The Aspire Needle will be utilized to extract the bone marrow and the Emcyte PureBMC will be used to concentrate bone marrow aspirate. The final concentrate will be injected into the hip.
  Arms: Bone marrow aspirate concentrate
Drug: Triamcinolone — 40 mg (1 mL) triamcinolone and 4 cc of lidocaine 1% that will be injected into the hip.
  Arms: Triamcinolone

SUMMARY:
This is a single site, randomized single blinded, two arm study researching the effects of bone marrow aspirate concentrate (BMAC) versus Triamcinolone in patients with hip osteoarthritis. The aims and hypothesis are as follows:

Specific Aim 1: Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months (6 weeks, 3 months, 6 months, and 12 months).

Hypothesis: The investigators hypothesize that triamcinolone and BMAC groups will have pain reduction after each respective intervention. The changes with triamcinolone will be noticeable on the short term. The BMAC changes will take longer to have an effect but will longer duration. The investigators hypothesize that at 6 months and 1 year participants receiving BMAC will have better scores reported on the WOMAC compared to the triamcinolone injection and better than prior to injection.

Specific Aim 2: Evaluate the change of bone marrow aspirate injection in comparison to triamcinolone in participant's performance on the 6 minute walk test from baseline to 12 months (6 weeks, 3 months, 6 months, and 12 months).

Hypothesis: The investigators hypothesize that there will be higher walking distances on the 6 minute walk test in the participants receiving a BMAC injection in comparison to triamcinolone starting at the 3 months follow-up time.

Specific Aim 3: Quantify and correlate cell characterization with patient reported outcomes score.

Hypothesis: The investigators hypothesize that there will be better patient reported outcomes in patients who have a higher concentration of mesenchymal stem cells injected.

The investigators will enroll 50 patients into each arm. Bone marrow will be aspirated then subsequently concentrated using the Emcyte PureBMC kit. The investigators will test the BMAC viability, rapid sterility, endotoxin, platelet concentration, volume, and total nucleated cell counts prior to injecting. The BMAC will be utilized as a hip injection into the affected hip of the patient.

Patients receiving the Triamcinolone will undergo a sham bone needling to simulate the aspiration to keep patients blinded. Both groups will receive their injections under ultrasound guidance.

DETAILED DESCRIPTION:
The goal of the study is to enroll 50 subjects in the bone marrow arm (BMAC group) and 50 in the triamcinolone arm (triamcinolone group). Once part fulfill the inclusion criteria, participants will be randomized to either intervention.

Participants will be enrolled in a staggering manner for the BMAC arm. The first 4 participants will be enrolled with at least 1 week interval in between these patients. During these weeks, the investigators will obtain results from the BMAC culture and evaluate safety response to the procedure. Participants enrolled in the triamcinolone arm will not be enrolled in a staggering manner, as the safety and efficacy are established as this is part of standard of care for hip osteoarthritis.

Participants will have the study protocol explained to them and will consent to the study, agreeing to have the bone marrow aspiration (BMA) and hip injection performed. Prior to any interventions, the participants will complete the baseline patient reported outcomes scores, and blood draw outlined in SOA section 1.3

Inclusion and exclusion criteria will be assessed during screening. Kellgren-Lawrence grade will be determined by blinded radiologists and co-investigators (Drs. Amer Hanano and Carl Winalski). An average score will be taken.

In order to blind the patient of the intervention, the triamcinolone group will undergo a "sham" bone needling of the bone cortex to simulate bone marrow harvesting (BMH). The posterior iliac spine will be anesthetized and needled simulating a BMH. Following the needling, the group will then receive a triamcinolone injection.

The process of aspirating the bone marrow used has been described by Dr. Friedlis and Dr. Centeno and will be completed under ultrasound guidance and in sterile fashion19. Multiple small draws of maximum 10 cc will be completed from different locations in the posterior superior iliac spine. The procedure as described is safe and been completed in more than 2000 individuals. Three to six passes are completed on each posterior superior iliac spine and a total volume of 60 cc of bone marrow is aspirated.

The BMAC group will have bone marrow aspirated using the Emcyte ASPIRE™ needle and subsequently concentrated using the Emcyte PureBMC™ system. Out of the bone aspirated, 60 cc will be utilized for concentration, 2 cc will be utilized by Bioscience Research Laboratory (BSR), and 2 cc will be stored in a -80°C biorepository enzyme-linked immunosorbent assay to determine concentrations of IL-1ra and other cytokines.

The 60 cc of unconcentrated bone marrow will then be concentrated to a total of 8 cc of concentrated bone marrow utilizing the Emcyte PureBMC™ system. Out of these 8 cc, 5 will be injected to the patient and the remainder 3 cc will be utilized for analyses.

These are the volumes and respective analyses:

* 1.5 cc will be directed to BSR for colony forming units, cell viability, total nucleated cell count as outlined in the subsequent paragaphs,
* 1 cc will be sent for 14 day culture
* 0.5 cc for endotoxin testing and gram stain

We will measure endotoxin concentrations utilizing the Charles River Nexgen PTS point of care instrument. The limit of endotoxin for general medical devices is 0.5 EU/mL. We will abide by this limit.

Rapid sterility will be assessed using a gram stain, performed by a CLIA certified laboratory at Cleveland Clinic Florida.

To ensure patient safety, patient will be considered a screen failure if there is a positive Gram stain or positive endotoxin testing. The injection of the BMAC will not be subsequently injected.

The remaining 5 cc will be utilized as the intervention group injectate. The BMAC will be injected as is and will not undergo any manipulation and/or dilution.

The 5 cc BMAC dose or 1 cc triamcinolone of 40 mg with 4 cc of lidocaine 1% will be injected into a single affected hip joint under ultrasound guidance.

Once the injection has been completed, patient will be monitored for 15 minutes and discharged home. Participants will be instructed to not use ice or anti-inflammatory medications for at least 6 weeks. For pain control following the procedure, the participant will be recommended to use acetaminophen or tramadol depending on the severity. Heat may be applied to the hip joint in case of muscle tightness. Ice should be avoided at the injection site. It may be applied at the site of bone marrow aspiration.

Participant will then follow-up in 6 weeks, 3 months, 6 months, and 1 year post-procedure to completed PROs and functional assessment with research staff. Participants will be asked to communicate to the Principal Investigator when anti-inflammatory medications are initiated, if necessary. Following the injections, both groups will resume home exercise program which participants had been completing prior to the injection in a pain free approach.

ELIGIBILITY:
Inclusion:

1. Provision of signed and dated consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged between 18 - 75 years old
4. WOMAC Pain Subscale With Average Score(Total WOMAC Pain Score Divided by 5) Equal to 4 or higher
5. Kellgren-Lawrence Grade greater than or equal to 2 on Hip X-Rays
6. Body Mass Index less than or equal to 35 kg/m2
7. Unilateral or Bilateral Hip Osteoarthritis
8. Prior physical therapy treatment for 6 weeks in the last 6 months
9. Agreement to adhere to Lifestyle Considerations (see section 5.3)
10. Discontinuation of pain/anti-inflammatory medications 2 week prior to baseline measurements
11. Patients with cancer in remission for at least 5 years. Specific cancers which were treated with surgical resection and are not undergoing chemotherapy/radiation therapy such as breast cancer, colon cancer, or skin cancer, and others could participate when deemed in remission for 1 year. Written approval from oncologist will be necessary prior to enrollment
12. Endotoxin less than or equal to 0.5 EU/ml
13. Negative gram stain result

Exclusion:

1. Prior corticosteroid injection to the hip
2. History of hip replacement(s)
3. Noncompliance to preventive screening tests for cancer indicated by age
4. Active autoimmune disease
5. Current use of oral corticosteroid
6. Use of immunosuppressive medications, or who are known to me immunocompromised
7. Inability to be weaned of oral anti-inflammatory medications
8. History of Diabetes or HbA1c > 6.5%
9. Uncontrolled Thyroid Dysfunction: 0.450 uIU/mL ≥ TSH levels ≥ 4.500 uIU/mL
10. Vitamin D Level < 30 ng/ml
11. Anemia (Hgb < 11.7 g/dL for Women; Hgb < 13 g/dL for men)
12. eGFR < 60 mL/min/1.73 m2
13. Thrombocytopenia with platelet count less than 150,000 x 109 L
14. Patients with coagulopathies based on known clotting disorder
15. Patients currently on anti-coagulation therapies
16. Patients who report any active infection(s) including cellulitis, TB, HIV, COVID, Hepatitis B and C
17. Moving over the next year
18. Inability to consent to the research study
19. Inability to complete forms electronically
20. Subjects in any other clinical trials
21. History of allergic reaction to lidocaine
22. Pregnancy or planning to be pregnant during trial
23. Breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Western Ontario McMaster Universities Arthritis Index (WOMAC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  WOMAC Scores range from 0 to 96, with higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario McMaster Universities Arthritis Index (WOMAC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  WOMAC Scores range from 0 to 96, with higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario McMaster Universities Arthritis Index (WOMAC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  WOMAC Scores range from 0 to 96, with higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Western Ontario McMaster Universities Arthritis Index (WOMAC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  WOMAC Scores range from 0 to 96, with higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  This outcome is used to measure the farthest distance walked within 6 minutes.
6 Minute Walk Test (6MWT) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  This outcome is used to measure the farthest distance walked within 6 minutes.
6 Minute Walk Test (6MWT) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  This outcome is used to measure the farthest distance walked within 6 minutes.
6 Minute Walk Test (6MWT) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  This outcome is used to measure the farthest distance walked within 6 minutes.

OTHER OUTCOMES:
PROMIS - Physical Function (PROMIS-PF) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Physical Function (PROMIS-PF) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Physical Function (PROMIS-PF) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Physical Function (PROMIS-PF) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Pain Interference (PROMIS-PI) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Pain Interference (PROMIS-PI) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Pain Interference (PROMIS-PI) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
PROMIS - Pain Interference (PROMIS-PI) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  All PROMIS instruments are calibrated to a mean t-score of 50 with a standard deviation of 10, with greater scores indicating more of the health domain in question (i.e., higher PROMIS-PF scores indicate greater function, whereas higher PROMIS-PI scores indicate that pain has a greater detriment on quality of life)
Global Rate of Change (GRoC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  GRoC range from -7 to 7 with lower scores indicating worse change.
Global Rate of Change (GRoC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  GRoC range from -7 to 7 with lower scores indicating worse change.
Global Rate of Change (GRoC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  GRoC range from -7 to 7 with lower scores indicating worse change.
Global Rate of Change (GRoC) | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  GRoC range from -7 to 7 with lower scores indicating worse change.
Pittsburgh Sleep Quality Index | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 weeks.
  The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.
Pittsburgh Sleep Quality Index | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 3 months.
  The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.
Pittsburgh Sleep Quality Index | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 6 months.
  The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.
Pittsburgh Sleep Quality Index | Evaluate the change in pain and functional scores of a single bone marrow aspirate injection in comparison to triamcinolone in patients with hip osteoarthritis through validated patient reported outcomes scores at baseline to 12 months.
  The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: LEONARDO P OLIVEIRA, MD, Principal Investigator — Cleveland Clinic Florida; Carlos Higuera-Rueda, MD, Study Director — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Hootman JM, Helmick CG, Barbour KE, Theis KA, Boring MA. Updated Projected Prevalence of Self-Reported Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation Among US Adults, 2015-2040. Arthritis Rheumatol. 2016 Jul;68(7):1582-7. doi: 10.1002/art.39692. PMID 27015600
- [Background] Duclos M. Osteoarthritis, obesity and type 2 diabetes: The weight of waist circumference. Ann Phys Rehabil Med. 2016 Jun;59(3):157-160. doi: 10.1016/j.rehab.2016.04.002. Epub 2016 May 19. PMID 27211819
- [Background] Courties A, Sellam J. Osteoarthritis and type 2 diabetes mellitus: What are the links? Diabetes Res Clin Pract. 2016 Dec;122:198-206. doi: 10.1016/j.diabres.2016.10.021. Epub 2016 Nov 5. PMID 27889689
- [Background] Quinn RH, Murray J, Pezold R, Hall Q. Management of Osteoarthritis of the Hip. J Am Acad Orthop Surg. 2018 Oct 15;26(20):e434-e436. doi: 10.5435/JAAOS-D-18-00351. PMID 30134309
- [Background] Kruse DW. Intraarticular cortisone injection for osteoarthritis of the hip. Is it effective? Is it safe? Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):227-33. doi: 10.1007/s12178-008-9029-0. PMID 19468910
- [Background] Hashmi SK. Basics of Hematopoietic Cell Transplantation for Primary Care Physicians and Internists. Prim Care. 2016 Dec;43(4):693-701. doi: 10.1016/j.pop.2016.07.003. PMID 27866586
- [Background] Charlesworth J, Fitzpatrick J, Perera NKP, Orchard J. Osteoarthritis- a systematic review of long-term safety implications for osteoarthritis of the knee. BMC Musculoskelet Disord. 2019 Apr 9;20(1):151. doi: 10.1186/s12891-019-2525-0. PMID 30961569
- [Background] Walters MC. Update of hematopoietic cell transplantation for sickle cell disease. Curr Opin Hematol. 2015 May;22(3):227-33. doi: 10.1097/MOH.0000000000000136. PMID 25767957
- [Background] Kim GB, Seo MS, Park WT, Lee GW. Bone Marrow Aspirate Concentrate: Its Uses in Osteoarthritis. Int J Mol Sci. 2020 May 2;21(9):3224. doi: 10.3390/ijms21093224. PMID 32370163
- [Background] Shapiro SA, Kazmerchak SE, Heckman MG, Zubair AC, O'Connor MI. A Prospective, Single-Blind, Placebo-Controlled Trial of Bone Marrow Aspirate Concentrate for Knee Osteoarthritis. Am J Sports Med. 2017 Jan;45(1):82-90. doi: 10.1177/0363546516662455. Epub 2016 Sep 30. PMID 27566242
- [Background] Rodriguez-Fontan F, Piuzzi NS, Kraeutler MJ, Pascual-Garrido C. Early Clinical Outcomes of Intra-Articular Injections of Bone Marrow Aspirate Concentrate for the Treatment of Early Osteoarthritis of the Hip and Knee: A Cohort Study. PM R. 2018 Dec;10(12):1353-1359. doi: 10.1016/j.pmrj.2018.05.016. Epub 2018 May 29. PMID 29857166
- [Background] Emadedin M, Ghorbani Liastani M, Fazeli R, Mohseni F, Moghadasali R, Mardpour S, Hosseini SE, Niknejadi M, Moeininia F, Aghahossein Fanni A, Baghban Eslaminejhad R, Vosough Dizaji A, Labibzadeh N, Mirazimi Bafghi A, Baharvand H, Aghdami N. Long-Term Follow-up of Intra-articular Injection of Autologous Mesenchymal Stem Cells in Patients with Knee, Ankle, or Hip Osteoarthritis. Arch Iran Med. 2015 Jun;18(6):336-44. PMID 26058927
- [Background] McIntyre JA, Jones IA, Han B, Vangsness CT Jr. Intra-articular Mesenchymal Stem Cell Therapy for the Human Joint: A Systematic Review. Am J Sports Med. 2018 Dec;46(14):3550-3563. doi: 10.1177/0363546517735844. Epub 2017 Nov 3. PMID 29099618
- [Background] Hernigou P, Trousselier M, Roubineau F, Bouthors C, Chevallier N, Rouard H, Flouzat-Lachaniette CH. Stem Cell Therapy for the Treatment of Hip Osteonecrosis: A 30-Year Review of Progress. Clin Orthop Surg. 2016 Mar;8(1):1-8. doi: 10.4055/cios.2016.8.1.1. Epub 2016 Feb 13. PMID 26929793
- [Background] Centeno CJ, Al-Sayegh H, Freeman MD, Smith J, Murrell WD, Bubnov R. A multi-center analysis of adverse events among two thousand, three hundred and seventy two adult patients undergoing adult autologous stem cell therapy for orthopaedic conditions. Int Orthop. 2016 Aug;40(8):1755-1765. doi: 10.1007/s00264-016-3162-y. Epub 2016 Mar 30. PMID 27026621
- [Background] Centeno CJ, Al-Sayegh H, Bashir J, Goodyear S, Freeman MD. A dose response analysis of a specific bone marrow concentrate treatment protocol for knee osteoarthritis. BMC Musculoskelet Disord. 2015 Sep 18;16:258. doi: 10.1186/s12891-015-0714-z. PMID 26385099
- [Background] Piuzzi NS, Mantripragada VP, Sumski A, Selvam S, Boehm C, Muschler GF. Bone Marrow-Derived Cellular Therapies in Orthopaedics: Part I: Recommendations for Bone Marrow Aspiration Technique and Safety. JBJS Rev. 2018 Nov;6(11):e4. doi: 10.2106/JBJS.RVW.18.00007. No abstract available. PMID 30461435
- [Background] Friedlis MF, Centeno CJ. Performing a Better Bone Marrow Aspiration. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):919-939. doi: 10.1016/j.pmr.2016.06.009. PMID 27788908
- [Background] Rezende MU, Gurgel HMC, Ocampos GP, Campos GC, Frucchi R, Pailo AF, Pasqualin T, Vicente JRN, Camargo OP. IMPROVEMENTS IN HIP OSTEOARTHRITIS WITH LAVAGE, TRIAMCINOLONE AND HYLAN G-F20. Acta Ortop Bras. 2020 Nov-Dec;28(6):280-286. doi: 10.1590/1413-785220202806240075. PMID 33328783
- [Background] Skwara A, Ponelis R, Tibesku CO, Rosenbaum D, Fuchs-Winkelmann S. Gait patterns after intraarticular treatment of patients with osteoarthritis of the knee--hyaluronan versus triamcinolone: a prospective, randomized, doubleblind, monocentric study. Eur J Med Res. 2009 Apr 16;14(4):157-64. doi: 10.1186/2047-783x-14-4-157. PMID 19380288
- [Background] Martin RL, Philippon MJ. Evidence of reliability and responsiveness for the hip outcome score. Arthroscopy. 2008 Jun;24(6):676-82. doi: 10.1016/j.arthro.2007.12.011. Epub 2008 Mar 12. PMID 18514111